CLINICAL TRIAL: NCT04454463
Title: Nonalcoholic Fatty Liver Disease (NAFLD) Database 3
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Baylor College of Medicine (Other); Case Western Reserve University (Other); Duke University (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Indiana University (Other); Liver Institute Northwest (Unknown); Seattle Children's Hospital (Other); St. Louis University (Other); University of California, San Diego (Other); University of California, San Francisco (Other); University of Southern California (Other); Virginia Commonwealth University (Other); Emory University (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: NAFLD Database 3; U01DK061732 (NIH); U01DK061713 (NIH); U01DK061737 (NIH); U01DK061718 (NIH); U01DK061734 (NIH); U01DK061738 (NIH); U01DK061728 (NIH); U01DK061731 (NIH); U24DK061730 (NIH); IRB00242326 (Other: JHM IRB)
Record Dates: First submitted 2020-06-05; First posted 2020-07-01 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Liver Diseases
Keywords: NAFLD; NASH; non-alcoholic steatohepatitis; fatty liver disease
MeSH Terms: conditions — Liver Diseases; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum, liver tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult patients with NAFLD: 1500 patients 18 years and older at the time of enrollment.
- Pediatric patients with NAFLD: 750 patients 2 years or older and up to 17 years old at the time of enrollment.

SUMMARY:
The NAFLD Database 3 will enroll approximately 1500 adult patients and 750 pediatric patients suspected or known to have NAFLD or NASH-related cirrhosis. To elucidate, through the cooperative effort of a multidisciplinary and multicenter group of collaborators, the etiology, natural history, diagnosis, treatment, and prevention of NAFLD, and in particular its more severe form of NASH and its complications.

DETAILED DESCRIPTION:
This is a multicenter, prospective follow-up study of patients with known nonalcoholic fatty liver disease (NAFLD) or nonalcoholic steatohepatitis (NASH). The primary objective of the study is to investigate the etiology, pathogenesis, natural history, diagnosis, treatment, and prevention of NAFLD and NASH.

ELIGIBILITY:
Inclusion Criteria:

* 2 years of age or older as of the initial screening interview and provision of consent
* Willingness to participate in the study for 1 or more years
* Histologic evidence of NAFLD or NASH based upon a standard of care liver biopsy
* Collection of serum and plasma up to 90 days before or 4- 90 days after standard of care liver biopsy
* Absence of regular or excessive use of alcohol within 2 years prior to initial screening

Exclusion Criteria:

* Clinical or histological evidence of alcoholic liver disease: Regular and excessive use of alcohol within the 2 years prior to interview defined as alcohol intake greater than 14 drinks per week in a man or greater than 7 drinks per week in a woman. Approximately 10 g of alcohol equals one 'drink' unit. One unit equals 1 ounce of distilled spirits, one 12-oz beer, or one 4-oz glass of wine
* Total parenteral nutrition for more than 1 month within a 6-month period before baseline liver biopsy
* Short bowel syndrome
* History of gastric or jejunoileal bypass preceding the diagnosis of NAFLD. Bariatric surgery performed following enrollment is not exclusionary. Liver biopsies obtained during bariatric surgery cannot be used for enrollment because of the associated surgical or anesthetic acute changes and the weight loss efforts that precede bariatric surgery
* History of biliopancreatic diversion
* Evidence of advanced liver disease defined as a Child-Pugh-Turcotte score equal to or greater than 10
* Evidence of chronic hepatitis B as marked by the presence of HBsAg in serum (patients with isolated antibody to hepatitis B core antigen, anti-HBc total, are not excluded)
* Evidence of chronic hepatitis C as marked by the presence of anti-HCV or HCV RNA in serum
* Low alpha-1-antitrypsin level and ZZ phenotype (both determined at the discretion of the investigator)
* Wilson's disease
* Known glycogen storage disease
* Known dysbetalipoproteinemia
* Known phenotypic hemochromatosis (HII greater than 1.9 or removal of more than 4 g of iron by phlebotomy)
* Prominent bile duct injury (florid duct lesions or periductal sclerosis) or bile duct paucity
* Chronic cholestasis
* Vascular lesions (vasculitis, cardiac sclerosis, acute or chronic Budd-Chiari, hepatoportal sclerosis, peliosis)
* Iron overload greater than 3+
* Zones of confluent necrosis, infarction, massive or sub-massive, pan-acinar necrosis
* Multiple epithelioid granulomas
* Congenital hepatic fibrosis
* Polycystic liver disease
* Other metabolic or congenital liver disease
* Evidence of systemic infectious disease
* Known HIV positive
* Disseminated or advanced malignancy
* Concomitant severe underlying systemic illness that in the opinion of the investigator would interfere with completion of follow-up
* Active drug use or dependence that, in the opinion of the study investigator, would interfere with adherence to study requirements
* Any other condition, which in the opinion of the investigator would impede compliance or hinder completion of study
* Inability to complete the appropriate informed consent process

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be at least 2250 patients age 2 years or older with histologically confirmed NAFLD or NASH located in the United States:
  * 1500 patients 18 years and older at the time of enrollment.
  * 750 patients 2 years or older and up to 17 years old at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 1649 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Change in alanine aminotransferase (ALT) levels from baseline to one year. | Baseline and 1 year
  ALT measure in IU/L (higher ALT indicates worse outcomes)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Sanyal, MD, Principal Investigator — Virginia Commonwealth University Medical Center; Brent Tetri, MD, Principal Investigator — St Louis University Hospital
Locations (16):
- United States (16):
  - University of California, San Diego- Adults, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California, San Diego Pediatrics, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Emory University-Pediatrics, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University- Adults, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - St. Louis University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Texas Children's Hospital, Baylor University, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Liver Institute Northwest, Seattle, Washington
  - Seattle Children's Hospital- SEA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The NASH CRN is fully committed to resource sharing beyond the NASH CRN investigators. The NASH CRN will make deposits to the NIDDK Central Data Repository according to the requirements outlined in the NIDDK Data Sharing Policy published in July 2013.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Within two years of end of the funding cycle.
Access Criteria: All qualified investigators will be allowed access to the stored materials at the end of a pre-determined proprietary period.
URL: https://repository.niddk.nih.gov/home

REFERENCES:
- See also: Nonalcoholic Steatohepatitis Clinical Research Consortium — http://jhuccs1.us/nash/
- See also: NIDDK Central Repository — https://repository.niddk.nih.gov/home